CLINICAL TRIAL: NCT03815552
Title: An Investigator Initiated Pilot Study to Evaluate the Impact on Glucose Control and Safety of the Eversense Continuous Glucose Monitoring System in Children and Adolescents
Brief Title: Evaluation of the Eversense Continuous Glucose Monitoring System in Type I Diabetic Youth
Acronym: FNH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kinderkrankenhaus auf der Bult (Other)
Collaborators: Senseonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-FNH-01
Record Dates: First submitted 2019-01-21; First posted 2019-01-24 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Self Care
Keywords: type 1 diabetes; pediatrics; blood sugar devices
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Eversense Continuous Glucose Monitoring (Experimental): The Eversense Continuous Glucose Monitoring System is a glucose monitoring device intended to continually measure interstitial fluid glucose levels in individuals with type 1 Diabetes.The System will be set to provide realtime glucose information, including alarms and alerts in the home settings für 180 days.
  Interventions: Device: Eversense Continuous Glucose Monitoring

INTERVENTIONS:
Device: Eversense Continuous Glucose Monitoring — The Eversense Continuous Glucose Monitoring System is a glucose monitoring device intended to continually measure interstitial fluid glucose levels in individuals with diabetes for the operating life of the sensor.The System comprises a sensor and a transmitter. The small sensor will be subcutaneously inserted in the arm.The transmitter reads glucose data from the subcutaneous sensor.
  Other Names: Senseonics Continuous Glucose Monitoring System

SUMMARY:
The purpose of this clinical investigation is to provide pilot clinical data to direct pivotal study development for the pediatric indication of the Senseonics Continuous Glucose Monitoring System (CGM) measurements when compared with finger stick blood glucose monitoring in an outpatient setting. (The investigation will also evaluate safety of the Senseonics CGM System usage, get feedback regarding subject and caregiver acceptability of the device and the mobile medical application (MMA).

DETAILED DESCRIPTION:
This is a non-randomized, non-blinded, prospective, single-arm, single-center pilot study, enrolling up to 15 pediatric subjects in two cohorts (5 subjects age 6-12 and 10 subjects age 13-17) with diabetes mellitus for up to 180 days. Study will evaluate the system at home with comparison to SMBG with clinic check visits and downloading of stored data every 30 days. Subjects will have one Sensor inserted subcutaneous by trained Investigators. The System will be set to provide real-time glucose information, including alarms and alerts in the home settings. The system is for adjunctive use. All diabetes care decisions will be based on SMBG values rather than System CGM results.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric subjects ≥6 and < 18 years with Type 1 Diabetes
2. HbA1c < 11 % at Screening
3. Subject/legal guardian has signed an informed consent form before any study related activities and is willing to comply with protocol requirements
4. Clinically confirmed diagnosis of diabetes mellitus for ≥ 1 year
5. Pretreated with CSII or ICT with a minimum duration of 3 month
6. Patient and parents are physically and mental able to exercise as determined the "Eversense" System
7. Patient must be willing to document every diabetes relevant information (meals, carbs, physical activity, extraordinary stress,…)
8. Patient is willing to follow protocol and procedures for study
9. Patient has the possibility to use a smartphone which is compatible with the system in daily life

Exclusion Criteria:

1. Patients are unwilling to follow the study procedures
2. Patient is absent for a longer time (no possibility for visits)
3. Patient is unable to tolerate tape adhesive in the area of sensor placement
4. Patient has any unresolved adverse skin condition in the area of sensor placement (e.g. atopic dermatitis, psoriasis, rash,…)
5. Patient is allergic to components of sensor material (Polymethylmethacrylate, dexamethasone, local anesthesia)
6. Eating disorder: e.g. bulimia, anorexia
7. Infections with hepatitis B, C or HIV
8. Coagulation disorder, wound healing disorder
9. Pregnancy
10. Mental incapacity or psychiatric disorders (Major Depression, anxiety disorders, schizophrenia)
11. Language barriers
12. Medication which is influencing metabolic control as systemic steroids, other non-Routine hormones
13. Medication influencing coagulation as Marcumar or systemic Xa-Antagonists as well as known bleeding disorders
14. People known to M. Addison
15. Untreated coeliac disease (Transglutaminase at screening elevated 2x>upper limit)
16. Severe diseases as cancer, heart failure, M. Parkinson, diabetic nephropathy or neuropathy or cardiomyopathy
17. Severe hypoglycemia in the past 3 months (defined as seizure or loss of consciousness)
18. Alcohol or drug abuse other than nicotine
19. Precluding adequate understanding or cooperation
20. A condition requiring or likely to require magnetic resonance imaging (MRI) during the study duration.
21. Any condition that in the investigator's opinion would make the subject unable to complete the study
22. Participation in another clinical investigation within 30 days or intent to participate during the study period
23. Patients with Diabetes mellitus Type 2.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
time in range | 90 days
  Reduction of time in range of Glucose < 70-mg/dL when using the Senseonics CGM System

SECONDARY OUTCOMES:
time of hypoglycemia | three weeks of the blinded phase compared to the last three weeks before 90 days visit
  Percentage time of hypoglycemia (Glucose <70 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Danne, MD, Study Chair — Kinder- und Jugendkrankenhaus AUF DER BULT
Locations (1):
- Kinder- und Jugendkrankenhaus AUF DER BULT, Hanover, Lower Saxony, Germany